CLINICAL TRIAL: NCT04279015
Title: The Effect Of Kinesio Tape In Chronic Neck Pain: Randomise Controlled Study
Brief Title: The Effect Of Kinesio Tape In Chronic Neck Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, MİNE PEKESEN KURTÇA, PT, PhD. Head of Physiotherapy Program, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014SBE013
Record Dates: First submitted 2020-02-10; First posted 2020-02-20 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Chronic Neck Pain
Keywords: Neck Pain; Kinesio tape; Pain; Quality of Life
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Intervention Model Description: pretest-posttest control groups in randomized parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional rehabilitation treatment (Active Comparator): Conventional physiotherapy program, consisting of standardised active (exercise) and passive (hotpack, ultrasound, conventional TENS) physical therapy methods, was applied by the same physiotherapist.
  Interventions: Procedure: Kinesio tape procedure
- Kinesio tape procedure (Active Comparator): In addition to the conventional physiotherapy program Kinesio tape was performed every day of conventional treatment immediately after the session ended by the same physiotherapist.
  Interventions: Procedure: Kinesio tape procedure

INTERVENTIONS:
Procedure: Kinesio tape procedure — Conventional rehabilitation treatment: Hotpack, ultrasound, conventional TENS and exercise for neck pain.
  Kinesio taping procedure: Inhibition technique with 15-25% tension to the upper trapezius muscle with I tape to reduce pain and muscle spasm, to support the weak muscles, Facilitation technique with Y-band with 15-35% tension to the cervical paravertebral muscles, and X-band with 15-35% tension to the rhomboideus major muscle technique and the correction technique was applied to the region where the individual defined the most pain and tenderness in palpation by using the "star application".
  Other Names: Conventional rehabilitation treatment

SUMMARY:
This study was planned to investigate the efficacy of treatment for Kinesio tape application in chronic neck pain individuals.

A total of 44 individuals were randomly divided into two groups (study group: 22, control group: 22). Conventional physiotherapy methods including active (exercise) and passive (hotpack, ultrasound and conventional transcutaneous electrical nerve stimulation (TENS)) treatment were applied to all subjects for 15 sessions (5 days a week). In addition to the individuals in the study group, Kinesio tape application was performed at the end of each session. Pain (Visual Analogue Scale), pressure pain threshold (digital algometer), range of motion (CROM device), muscle strength (Hand-Held Dynamometer), muscle endurance, pectoralis minor muscle length, quality of life (Nottingham Health Profile) and depressive symptoms (Beck Depression Scale) assessments were performed before treatment, on the second day of treatment and after treatment (after three weeks). Treatment satisfaction with individuals (Visual Analogue Scale) was assessed on the 2nd day of treatment and post-treatment (after three weeks).

DETAILED DESCRIPTION:
In the literature, it is seen that Kinesio tape is used in problems such as knee pain, chronic low back pain, neck pain, shoulder pain and common musculoskeletal pain. Some studies with individuals with low back and neck pain show positive effects of Kinesio tape on pain reduction and recovery in disability. However, studies are reporting the opposite of these results. The number of studies in the literature is insufficient to create clinical evidence regarding the use of Kinesio tape in patients with neck pain. By considering this deficiency, the purpose of our study was to investigate the effect of Kinesio tape applied together with conventional physiotherapy methods in individuals with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 30-55,
* Having been suffering from neck pain for at least three months,
* Getting at least 5 points from the Neck Disability Index,
* Having pain between the superior nuchal line and spina scapula,
* Neck Pain Task Force, which consists of four levels to be at the first and second level.

Exclusion Criteria:

* Presence of conditions that will prevent evaluation or communication (such as cognitive problems),
* Being illiterate,
* Having had physiotherapy from the neck, back or waist region in the last six months,
* Having had cervical region and spine surgery,
* Presence of impingement or thoracic outlet syndrome, malignancy, fractured, systemic autoimmune diseases, neurological problems and diagnosed psychiatric diseases that will prevent evaluation and treatment.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Evaluations were made before treatment, on the 2nd day of treatment and after 3 weeks (1 day after completion of treatment) by the same physiotherapist.
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.Visual Analogue Scale was used to evaluate pain intensity. The highest score is 10, the lowest is 0. High scores indicate that pain intensity is high.
Pressure pain threshold | Evaluations were made before treatment, on the 2nd day of treatment and after 3 weeks (1 day after completion of treatment) by the same physiotherapist.
  Pressure pain threshold was evaluated with an objective method, digital algometer. The results are recorded in Newton / cm2.
Cervical range of motion | Evaluations were made before treatment, on the 2nd day of treatment and after 3 weeks (1 day after completion of treatment) by the same physiotherapist.
  Cervical range of motion was evaluated with the Cervical Range of Motion device.All movements were actively carried out, and measurement results were recorded in degrees.
Isometric muscle strengths | Evaluations were made before treatment, on the 2nd day of treatment and after 3 weeks (1 day after completion of treatment) by the same physiotherapist.
  Isometric muscle strengths of the cervical region were evaluated by Hand-Held Dynamometer. The result measurements were recorded in Newton.
The pectoralis minor muscle shortness | Evaluations were made before treatment, on the 2nd day of treatment and after 3 weeks (1 day after completion of treatment) by the same physiotherapist.
  The pectoralis minor muscle shortness of the participants was evaluated with a standard bilateral ruler.Muscle shortness was recorded in centimetres.
The endurance of the deep neck flexor muscles | Evaluations were made before treatment, on the 2nd day of treatment and after 3 weeks (1 day after completion of treatment) by the same physiotherapist.
  The endurance of the deep neck flexor muscles with a chronometer, muscle endurance was recorded in seconds.

SECONDARY OUTCOMES:
Neck Disability Index | Evaluations were made before treatment, on the 2nd day of treatment and after 3 weeks (1 day after completion of treatment) by the same physiotherapist.
  Disability levels of the participants were assessed with the Neck Disability Index.The highest score is 50, the lowest is 0. High scores indicate that disability level is high.
Nottingham Health Profile | Evaluations were made before treatment, on the 2nd day of treatment and after 3 weeks (1 day after completion of treatment) by the same physiotherapist.
  Quality of life were assessed with Nottingham Health Profile.The highest score is 600, the lowest is 0. The increase in score indicates worse quality of life.
Beck Depression Inventory | Evaluations were made before treatment, on the 2nd day of treatment and after 3 weeks (1 day after completion of treatment) by the same physiotherapist.
  The emotional status were assessed with Beck Depression Inventory. The highest score that can be obtained is 63, the lowest is 0. It has been reported that individuals scoring 17 points or more have severe depressive symptoms that require treatment.
Treatment satisfaction | Evaluations were made on the 2nd day of treatment and after 3 weeks (1 day after completion of treatment) by the same physiotherapist.
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.Treatment satisfaction were assessed with the Visual Analogue Scale. The highest score is 10, the lowest is 0. High scores indicate that treatment satisfaction is high.

IPD SHARING:
Plan to Share IPD: No